CLINICAL TRIAL: NCT07040306
Title: A Prospective Clinical Follow-up Study of Drug Treatment in Patients With Graves' Disease
Brief Title: A Clinical Follow-up Study on Drug Therapy for Graves' Disease Patients in China
Status: Recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Xiaochun Teng, Chief Physician, First Hospital of China Medical University
Other Study IDs: 2019-222
Record Dates: First submitted 2025-06-03; First posted 2025-06-27 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Graves´ Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Save blood samples (whole blood and serum) of enrolled GD patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Methimazole(MMI) — Determine the enrolled GD patients and adjust the dosage of methimazole according to the 2016 American Thyroid Association guidelines. Conduct thyroid function, liver function, TRAb, and blood routine tests during outpatient follow-up to observe the treatment effect and provide medication guidance.

SUMMARY:
This study was a prospective follow-up study of newly diagnosed and relapsed Graves' disease patients in the Endocrinology Clinic of the First Affiliated Hospital of China Medical University. The following aspects will be studied: 1. Through the prospective follow-up study of GD patients, we will get the relapse rate and remission rate of GD patients treated with drugs, explore the risk factors of GD patients relapsing after drug treatment, and make GD relapse risk prediction software; 2. To compare the effects of high dose and low dose methimazole on the remission rate, liver side effects, leukopenia and other adverse drug reactions, and to summarize the incidence and risk factors of liver side effects, leukopenia and other adverse drug reactions caused by drug treatment; 3. To investigate the sensitivity and specificity of TRAb in the diagnosis of GD in China and its role in predicting recurrence; 4. After taking ATD, the serum alkaline phosphatase of GD patients will increase first and then decrease. This study will focus on analyzing the dynamic changes of this index before and after methimazole treatment, and analyze the relationship between it and thyroid function index.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Newly diagnosed GD and GD relapses.

Exclusion Criteria:

1. Patients with active infiltrative exophthalmos in GD were excluded.
2. Patients with other autoimmune diseases affecting thyroid function were excluded.
3. Excluding patients with combined malignancies and other serious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population includes male and female hyperthyroidism patients over the age of 18. Participants must have no history of autoimmune hepatitis, viral hepatitis, blood disease, bone marrow or liver transplantation, and complete clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-11-14 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Relapse and remission of Graves' disease in adult treated with methimazole. | 30 years
  Relapse was defined as having clinical and biochemical hyperthyroidism (FT3 and FT4 increased and TSH decreased) after discontinuation of methimazole. Remission is defined as having clinical and biochemical euthyroidism(FT3, FT4 and TSH are normal) without methimazole treatment for at least 12 months. Through the prospective follow-up study of GD patients, we will get the relapse rate and remission rate of GD patients treated with drugs, explore the risk factors of GD patients relapsing after drug treatment, and make GD relapse risk prediction software.
Adverse effects of methimazole in the treatment of Graves' disease in adult. | 30 years
  Adverse effects are defined as having neutropenia (absolute neutrophil count< 1800/µL), liver dysfunction (AST or ALT> 60 IU/L), rash, arthralgia, myalgia, et al. To compare the effects of high dose and low dose methimazole on the remission rate, liver side effects, leukopenia and other adverse drug reactions, and to summarize the incidence and risk factors of liver side effects, leukopenia and other adverse drug reactions caused by drug treatment

SECONDARY OUTCOMES:
Thyrotropin receptor antibody(TRAb) | 30 years
  To investigate the sensitivity and specificity of the thyrotropin receptor antibody(TRAb) in the diagnosis of GD in China and its role in predicting recurrence
The serum alkaline phosphatase | 30 years
  After taking ATD, the serum alkaline phosphatase of GD patients will increase first and then decrease. This study will focus on analyzing the dynamic changes of this index before and after methimazole treatment, and analyze the relationship between it and thyroid function index

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT07040306/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT07040306/ICF_002.pdf